CLINICAL TRIAL: NCT00851396
Title: Assessment of Influence of Vitamin D on Insulin Secretion and Sensitivity in Obese Teenage Girls (Assessment of Prevalence of Vitamin D Deficiency in Obese Teenage Girls and Influence of Vitamin D on Insulin Secretion and Sensitivity)
Brief Title: Assessment of Influence of Vitamin D on Insulin Secretion and Sensitivity in Obese Teenage Girls
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ambika Ashraf, M.D., Assistant Professor, Pediatrics, University of Alabama at Birmingham
Other Study IDs: F080221001
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Vitamin D Deficiency; Insulin Resistance; Insulin Sensitivity; Obesity
Keywords: Vitamin D deficiency; Insulin resistance; Glucose- Insulin dynamics; Obese adolescents
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese female adolescents: Obese adolescents will be screened for vitamin D deficiency through an existing study. Those found to be vitamin D deficient will be given standard treatment of vitamin D deficiency. In this study, patients who self report that they had taken the treatment for vitamin D will be screened for serum 25 OH D level and will undergo OGTT. The OGTT results as well as insulin resistance indices will be compared to their initial values.

SUMMARY:
The purpose of the study is to assess the relationship between vitamin D status and insulin- glucose dynamics in obese Adolescents. The study is intended to assess the difference in the insulin sensitivity before and after correction of vitamin D deficiency.

DETAILED DESCRIPTION:
The vitamin D deficient subjects are identified initially through an existing study. Those identified with vitamin D deficiency are notified and subsequently treated with standard therapy for vitamin D deficiency as part of their clinical care. Patients who self report that they have taken the treatment are enrolled in this study. Patients will be evaluated in this study with measurement of serum 25 OH D level, PTH and oral glucose tolerance test. The study will assess if there is improvement in glucose- insulin sensitivity dynamics once the serum 25OH D level is normalized

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents who are menarchal
* BMI is 95th centile, for age and sex
* Patients will be screened for vitamin D deficiency through an existing study.
* Those found to be vitamin D deficient will be given standard treatment of vitamin D deficiency.
* In this study, patients who self report that they had taken the treatment for vitamin D will be screened for serum 25 OH D level

Exclusion Criteria:

* Children with diabetes, other endocrine or acute or chronic medical illnesses, children on oral contraceptive pills, diuretics and anticonvulsant medications

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female adolescents who are menarchal BMI is 95th centile, for age and sex
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The insulin secretory capacity and insulin resistance indices are the outcome of interest in this study. | December 2009

SECONDARY OUTCOMES:
We will evaluate whether the relationship of obesity and insulin resistance and the defective insulin secretory capacity is modulated by vitamin D status | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital , University of Alabama, Birmingham, Alabama, United States